CLINICAL TRIAL: NCT07377461
Title: Comparative Study of Access Sheaths With Flexible Tips and Suction Versus Conventional Access in Endourology: A Prospective Study
Brief Title: Flexible and Navigable Suction Ureteral Access Sheath (FANS) vs Conventional Access Sheaths in RIRS: A Prospective Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0069-24-BRZ
Record Dates: First submitted 2026-01-07; First posted 2026-01-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones; Nephrolithiasis
Keywords: Retrograde Intrarenal Surgery; Ureteral Access Sheath; Suction Ureteral Access Sheath; Flexible Tip Ureteral Access Sheath; RIRS; Operative Time; Endourology
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio to one of two parallel intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible and Navigable Suction Ureteral Access Sheath (FANS) (Experimental): Participants underwent retrograde intrarenal surgery using a flexible and navigable ureteral access sheath with integrated suction capability.
  Interventions: Device: Flexible and Navigable Suction Ureteral Access Sheath (FANS)
- Conventional Ureteral Access Sheath (Active Comparator): Participants underwent retrograde intrarenal surgery using a standard, non-suction ureteral access sheath.
  Interventions: Device: Conventional Ureteral Access Sheath

INTERVENTIONS:
Device: Flexible and Navigable Suction Ureteral Access Sheath (FANS) — Use of a flexible distal-tip ureteral access sheath with integrated suction during retrograde intrarenal surgery to facilitate access, irrigation control, and fragment evacuation.
  Arms: Flexible and Navigable Suction Ureteral Access Sheath (FANS)
Device: Conventional Ureteral Access Sheath — Use of a standard ureteral access sheath without suction during retrograde intrarenal surgery.
  Arms: Conventional Ureteral Access Sheath

SUMMARY:
Kidney stones located in the kidney are commonly treated using a minimally invasive procedure called retrograde intrarenal surgery (RIRS). During this procedure, a ureteral access sheath is often used to facilitate repeated access to the kidney, improve visualization, and allow irrigation fluid to drain.

Newer access sheaths have been developed with flexible distal tips and built-in suction capabilities, which may help reduce operative time by improving visibility and removing stone fragments and irrigation fluid more efficiently.

This prospective randomized study compared a flexible and navigable suction ureteral access sheath with a conventional ureteral access sheath in adult patients undergoing RIRS for kidney stones measuring 10 mm or larger. Participants were randomly assigned to one of the two access sheath types.

The primary objective of the study was to evaluate whether the use of a suction-enabled access sheath reduces operative time. Secondary objectives included assessment of complications, length of hospital stay, stone-free rate, and need for additional interventions.

DETAILED DESCRIPTION:
This was a prospective, single-center, randomized controlled trial conducted at a tertiary referral endourology center. Adult patients (≥18 years) with renal stones measuring 10 mm or greater and scheduled to undergo retrograde intrarenal surgery (RIRS) under general anesthesia were eligible for inclusion.

Participants were randomized in a 1:1 ratio to undergo RIRS using either a flexible and navigable suction ureteral access sheath (FANS group) or a conventional ureteral access sheath (control group). Randomization was performed using a computer-generated sequence with allocation concealment via sealed opaque envelopes. Blinding of the operating surgeon was not feasible due to the nature of the devices used.

All procedures were performed by experienced endourologists using standardized surgical techniques. Flexible ureteroscopy was performed with a digital ureteroscope, and stone fragmentation was achieved using a Holmium:YAG laser in dusting mode. In the suction access sheath group, negative pressure suction was applied through the sheath according to manufacturer guidelines. Irrigation parameters were standardized across both study arms.

The primary outcome measure was operative time, defined as the interval from insertion of the first endoscopic instrument through the urethra to removal of the final instrument at the end of the procedure. Secondary outcome measures included intraoperative and postoperative complications (classified using the Clavien-Dindo system), ureteral wall injury, length of hospital stay, stone migration, and stone-free rate. Stone-free status was defined as the absence of residual fragments greater than 2 mm on postoperative imaging.

Preoperative assessment included non-contrast computed tomography to evaluate stone size, location, and burden. Postoperative imaging was performed using kidney-ureter-bladder radiography or renal ultrasound approximately two weeks after surgery.

The study was approved by the Institutional Review Board of Barzilai University Medical Center, and all participants provided written informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Presence of single or multiple renal stones measuring 10 mm or greater

Eligible for retrograde intrarenal surgery under general anesthesia

Ability to provide written informed consent

Exclusion Criteria:

Pregnancy

Active urinary tract infection at the time of surgery

Known bleeding disorders

Solitary kidney

Anatomical abnormalities of the urinary tract that could affect ureteroscopic access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Operative Time | During the surgical procedure
  Operative time was defined as the duration from insertion of the first endoscopic instrument through the urethra to removal of the final instrument at the end of the procedure.

SECONDARY OUTCOMES:
Intraoperative and Postoperative Complications | Perioperative period (Day of surgery through postoperative Day 30).
  Intraoperative and postoperative complications were recorded and classified according to the Clavien-Dindo classification system.
Stone-Free Rate | Two weeks after surgery
  Stone-free status was defined as the absence of residual stone fragments greater than 2 mm on postoperative imaging.
Length of Hospital Stay | From end of surgery until hospital discharge (typically 1-3 days).
  Length of hospital stay was defined as the number of days from surgery to hospital discharge.
Ureteral Wall Injury | During the surgical procedure
  Ureteral wall injury was assessed intraoperatively and classified according to the Traxer-Thomas classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No